CLINICAL TRIAL: NCT05274308
Title: Cascadion™ SM Immunosuppressants Panel, Stability of Tacrolimus, Cyclosporine A, Everolimus and Sirolimus in Whole Blood Patient Samples
Brief Title: Stability of Tacrolimus, Cyclosporine A, Everolimus and Sirolimus in Whole Blood Patient Samples
Status: Completed | Type: Observational
Sponsor: Thermo Fisher Scientific Oy (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: CA1803-STSS-PRO
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Transplantation Drugs Stability
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples in K2 EDTA tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient blood sample collection: 30 mL of whole blood collected from eligible patients in one sampling
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling from all eligible transplantation patients according to the protocol

SUMMARY:
This is a prospective, observational evaluation study to assess the stability of the analytes tacrolimus, cyclosporine A, everolimus and sirolimus measured with Cascadion™ SM Immunosuppressants Panel. Study is pre-market evaluation for the regions where Cascadion™ SM Immunosuppressants Panel is not on the market yet and post-market evaluation where it is.

To assess the stability of tacrolimus, cyclosporine A, everolimus and sirolimus in patient whole blood samples after they are collected, processed and subjected to various storage conditions or freeze-thaw cycles that represent common sample handling conditions in the commercial clinical laboratory setting.

Study subjects will undergo one venous sample collection where 30 mL of blood is drawn.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Ability to sign informed consent form
3. At least one of the following

   1. Kidney, liver or heart transplant patient using tacrolimus or cyclosporine A
   2. Kidney or liver transplant patient using everolimus
   3. Kidney transplant patient using sirolimus

Exclusion Criteria:

1. Inability to provide informed consent
2. Pregnancy or breastfeeding
3. Likely to believe that the sample collection procedure will pose an unusually high risk for subject's physical or mental health or their comfort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject's using following immunosuppressants drugs accordingly with organ transplantation
  1. Kidney, liver or heart transplant patient using tacrolimus or cyclosporine A
  2. Kidney or liver transplant patient using everolimus
  3. Kidney transplant patient using sirolimus
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Acceptance criteria for claiming the patient samples storage stability | 5 months
  Stability of cyclosporine A, tacrolimus, everolimus and sirolimus in patient whole blood samples will be tested at +15-25°C up to 4 days, at +2-8°C up to 15 days and at -20±5°C up to 31 days. Relative bias at each time point to T0 baseline is calculated for each patient sample separately. The grand average relative bias across all samples, and the associated 95% confidence interval, must be within -15% and +15%.

CONTACTS AND LOCATIONS:
Overall Officials: Sanna Anttonen, Study Director — Thermo Fisher Scientific, Inc
Locations (1):
- AOU Città della Salute e della Scienza di Torino/S.C Biochimica Clinica, Turin, Italy

IPD SHARING:
Plan to Share IPD: No